CLINICAL TRIAL: NCT03293979
Title: Alere i FluA*B Biologic Test Relocated in Emergency Service for Flu Diagnosis
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: TestAiFluA&B
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Test A i Flu A&B implemented in emergency service — Test A i Flu A&B implemented in emergency service

SUMMARY:
It appears that the heavyness of flu pathology, the diagnosis limits and the validity of it was well studied in the last years.However, the economical impact and the organisation benefit in emergency service is not yet evaluated Our purpose is to study the impact of implementation of fast flu diagnosis by molecular biology available in emergency service in the economic field .

ELIGIBILITY:
Inclusion Criteria:

* respiratory symptoms
* fever >38°C
* general symptoms of flu like pathology

Exclusion Criteria:

* cognitive disorders
* patient with guardianship
* patient already having a flu diagnosis in the last 7 days
* without social protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: each patient admitted in emergy service between february 2016 and april 2016
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
time to have the result of the biological test | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: GANANSIA Olivier, MD, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No